CLINICAL TRIAL: NCT04002778
Title: Rapid On-Site Evaluation (ROSE) by Endosonographer: for Whom, When and by Whom?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Guilherme Rezende, Associate Professor, Internal Medicine, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 45073415.3.0000.5257
Record Dates: First submitted 2019-05-20; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Pancreatic Neoplasms
Keywords: EUS-FNA; pancreatic solid lesions; sample adequacy; cytopathology; endosonography
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROSE by endosonographer (Active Comparator): Submitted to fine-needle aspiration. Endosonographer's on-site evaluation of sample adequacy and categorization
  Interventions: Diagnostic Test: Fine needle aspiration; Diagnostic Test: Rapid on-site evaluation
- non-ROSE (Other): Submitted to fine-needle aspiration.
  Interventions: Diagnostic Test: Fine needle aspiration

INTERVENTIONS:
Diagnostic Test: Fine needle aspiration
Diagnostic Test: Rapid on-site evaluation
  Arms: ROSE by endosonographer

SUMMARY:
Endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA) is a highly sensitive and specific method in diagnosing solid pancreatic lesions. Rapid on-site evaluation (ROSE) of the aspirate by a cytopathologist improves specimen adequacy and diagnostic accuracy while reducing the number of needle passes. As this increases costs and implicates availability issues, the investigators aimed to evaluate the utility of ROSE by the endosonographer in guiding EUS-FNA of solid pancreatic lesions.

DETAILED DESCRIPTION:
Consecutive patients with a solid pancreatic lesion were included. Endosonographer was submitted to a basic pancreatic cythpatology training programme at two institutitions. The patients were randomly allocated to the ROSE group - in which the number of needle passes required to obtain a sample suitable for cytopathologic categorization was established by the endosonographer's on-site evaluation - or to the non-ROSE group - in whom adequacy of the specimen was evaluated macroscopically and up to five needle passes could be performed, assuring sample adequacy. The gold standard was the final cytopathologist's diagnosis. The number of needle passes, procedure duration, specimen adequacy, diagnostic yield and adverse events rates were compared between groups and the performance measures of ROSE by endosonographer were determined.

ELIGIBILITY:
Inclusion Criteria:

* solid pancreatic lesions detected by trans abdominal ultrasound or cross-sectional image (CT or MRI).
* formal indications to undergo EUS-FNA which were: differentiation between benign and malignant diseases, radiologic criteria of inoperability or unresectability, need for specific diagnosis which could modify therapeutic strategy and need for a diagnosis before neoadjuvant therapy.

Exclusion Criteria:

* a cystic or solid cystic aspect of the pancreatic lesion on above mentioned image methods
* lesions previously punctured on past EUS-FNA procedures
* American Society of Anesthesiologist (ASA) Physical Status Classification System IV or V
* cases of surveillance of solid pancreatic lesions
* severe coagulation disorder (platelet count < 50000 or International Normalized Ratio > 2,0)
* impossibility of previous suspension of antiplatelet agents (except acetylsalicylic acid) or anticoagulants (all)
* patient unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Procedure duration | Procedure
  Minutes

SECONDARY OUTCOMES:
Specimen adequacy rate | Through study completion, an average of 18 months
  Cases with a sample suitable for a definitive diagnosis over the total number of cases
Total number of passes | Through study completion, an average of 18 months
  total number of passes of all procedures
Number of adverse events | Through study completion, an average of 18 months
  Total number of adverse events of all procedures
Diagnostic yield | Through study completion, an average of 18 months
  Cases in which a final diagnostic could be established over the total number of cases

IPD SHARING:
Plan to Share IPD: Undecided